CLINICAL TRIAL: NCT05807932
Title: Phase-I/II Trial to Assess the Safety and Efficacy of Venetoclax in Addition to Sequential Conditioning With Fludarabine / Amsacrine / Ara-C (FLAMSA) + Treosulfan for Allogeneic Blood Stem Cell Transplantation in Patients With MDS, CMML or sAML (FLAMSAClax
Brief Title: Venetoclax in Addition to Sequential Conditioning With Fludarabine / Amsacrine / Ara-C (FLAMSA) + Treosulfan for Allogeneic Blood Stem Cell Transplantation in Patients With MDS, CMML or sAML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Koordinierungszentrum für Klinische Studien - Duesseldorf (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLAMSAClax
Record Dates: First submitted 2023-03-03; First posted 2023-04-11 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: MDS; sAML; CMML; allogeneic blood stem cell transplantation; Venetoclax
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — venetoclax; Amsacrine; Cytarabine; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax (Experimental): Venetoclax treatment will be started orally once a day with food, one day before FLAMSA conditioning therapy and stopped the day before high-dose Treosulfan. The total duration of treatment with Venetoclax will be 6 days (day -11 to -6 before stem cell infusion). Patients with active disease at transplant will receive a 3-day ramp-up prephase of Ara-C (100mg total dose infused in 1h) with daily increasing doses of Venetoclax to prevent TLS during conditioning. Total treatment duration with Venetoclax in patients with active disease at transplant will be 8 days (day -13 to -6 before stem cell infusion).
  Interventions: Drug: Venetoclax; Drug: Amsacrine; Drug: Ara-C; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Venetoclax — Study treatment consists of the conditioning therapy including 6 or 8 days of Venetoclax treatment.
Drug: Amsacrine — Amsacrine is part of the conditioning therapy and is administered on day -10 to -7 before allogeneic blood stem cell transplantation
Drug: Ara-C — Ara-C is part of the conditioning therapy and is administered on day -10 to -7 before allogeneic blood stem cell transplantation
Drug: Tacrolimus — Tacrolimus is used for prophylaxis of acute and chronic graft-versus-host-disease according to institutional standards.
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil is used for prophylaxis of acute and chronic graft-versus-host-disease according to institutional standards.

SUMMARY:
This trial aims to find the MTD of Venetoclax when added to Fludarabin, Amsacrine and Ara-C + Treosulfan and to evaluate whether the addition of Venetoclax to sequential conditioning with FLAMSA + Treosulfan is safe for allogeneic blood stem cell transplantation in patients with high-risk MDS, CMML or sAML (FLAMSAClax)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC), prior to the initiation of any study-specific procedures
* MDS, CMML or sAML according to WHO classification (revised version 2016) with a marrow blast count >5% and/or high-risk genetic features (e.g. bad risk karyotype according to the IPSS-R / ELN classification or presence of unfavorable somatic mutations (e.g. TP53, RUNX1, IDH1, IDH2, KMT2A, DEK-NUP214 or RAS pathway mutations including NRAS, KRAS, PTPN11, CBL, NF1, RIT1 or KIT), falling into the "high" or "very high" risk category of the IPSS-R or IPSS-M) any time between diagnosis and inclusion
* Untreated except for oral Hydroxyurea or a maximum of 2 courses of treatment with Azacytidine or Decitabine alone or in combination with Venetoclax
* Identification of a well matched (10 out of 10, A, B, C, DR, DQ) donor either related or unrelated
* Age ≥18
* HCT-CI ≤ 3 (except former treatment of a solid tumor)
* ECOG performance status ≤ 2 at study entry
* no active, uncontrolled infection at inclusion
* able to adhere to the study visit schedule and other protocol requirements
* Female of childbearing potential (FCBP) must:

  * Understand that based on embryo-foetal toxicity studies in animals venetoclax may harm the foetus when administered to pregnant woman
  * Agree to have a medically supervised pregnancy test at Screening and within 72 hours prior treatment start
  * Avoid becoming pregnant while receiving Venetoclax
  * Use effective contraception during treatment with Venetoclax and for at least 1 months after the last dose,
  * Understand that is currently unknown whether venetoclax may reduce the effectiveness of hormonal contraceptives, and therefore women using hormonal contraceptives should add a barrier method
  * Notify her study doctor immediately if there is a risk of pregnancy
* Males must:

  * agree to use condoms, even if the male subject has undergone a successful vasectomy, from Study Day 1 through at least 30 days after the last dose of study drug.
  * Agree to notify the investigator immediately, if pregnancy or a positive pregnancy test occurs in his partner during study participation

Exclusion Criteria:

* sAML with known FLT3 mutation (ITD or TKD)
* Marrow blast count >30% at the time of screening
* Peripheral white blood count >20,000 per microliter despite treatment with Hydroxyurea
* previous cytotoxic therapy exceeding oral Hydroxyurea or >2 courses of treatment with Azacytidine, Decitabine or low dose Ara-C alone or in combination with Venetoclax
* previous allogeneic blood stem cell transplantation
* symptomatic CNS-involvement with MDS; CMML or sAML
* any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* pregnant or lactating females
* Refusal to use safe contraceptive methods during the study period
* Cardiac history of CHF (>NYHA 2) requiring treatment or Ejection Fraction < 40% or chronic stable angina
* Forced expiratory volume in 1 second (FEV1) <50% of expected corrected for hemoglobin and/or volume
* Diffusing capacity of the lungs for carbon monoxide (DLCO) <50% of expected corrected for hemoglobin and/or volume
* any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study:

  * Impaired renal function (GFR < 45 ml/min)
  * Impaired hepatic function, as follows Aspartate aminotransferase (AST) ≥3 x ULN or Alanine aminotransferase (ALT) ≥3 x ULN or Total bilirubin ≥1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin) or Alkaline Phosphatase ≥3 x ULN
* known hypersensitivity to Venetoclax, Fludarabine, Amsacrine, Ara-C or Treosulfan
* concurrent use of other anti-cancer agents or treatments except Hydroxyurea and a maximum of 2 courses of Azacytidine or Decitabine
* positive for HIV or replicating infectious hepatitis, type A, B, C or E
* prior history of malignancy other than MDS, CMML, sAML (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 2 years
* participation in another study with ongoing use of unlicensed investigational product from 28 days or <5 half-lifes of the investigational product before study enrollment
* No planned or executed/given treatment with any of the following within 7 days prior to the first dose of study drug (or ramp-up prophase):

  * Steroid therapy for anti-neoplastic intent
  * moderate or strong cytochrome P450 3A (CYP3A) inhibitors
  * moderate or strong CYP3A inducers
* Refusal to avoid consumption of any of the following within 3 days prior to the first dose of study drug: grapefruit or grapefruit products, Seville oranges (including marmalade containing Seville oranges), star fruit.
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary target variable is safety, defined as the maximal organ toxicity to each organ system according to CTC criteria as well as the number of AEs of grade III or greater within the first 30 days (± 3) after transplantation | inclusion until day 30 (± 3) after transplantation
  maximal organ toxicity to each organ system according to CTC criteria as well as the number of AEs of grade III or greater within the first 30 days (± 3) after transplantation

SECONDARY OUTCOMES:
Safety, defined as the maximal organ toxicity to each organ system according to CTC criteria as well as the number of AEs of grade III or greater until day +100 (± 7) after transplantation | inclusion until day +100 (± 7) after transplantation
  maximal organ toxicity to each organ system according to CTC criteria as well as the number of AEs of grade III or greater until day +100 (± 7) after transplantation
Graft failure at day +30 (± 3) after transplantation | transplantation until day +30 (± 3) after transplantation
  Number of patients with graft failure (no donor chimerism at day +30 (± 3) after transplantation)
Incidence of aGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Incidence of aGvHD during the first 2 years after transplantation
Course of aGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Course of aGvHD during the first 2 years after transplantation (response/no response to steroids)
Severity of aGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Severity of aGvHD during the first 2 years after transplantation (according to Glucksberg criteria)
Incidence of cGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Incidence of cGvHD during the first 2 years after transplantation
Course of cGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Course of cGvHD during the first 2 years after transplantation (response/no response to steroids)
Severity of cGvHD during the first 2 years after transplantation | transplantation until 2 years after transplantation
  Severity of cGvHD during the first 2 years after transplantation (according to NIH criteria)
Incidence, course and severity of VOD | transplantation until 2 years after transplantation
  Incidence, course and severity of VOD (according to EBMT criteria)
Time to hematopoietic reconstitution | From date of transplantation (day 0) until the date of first documented hematopoietic reconstitution, assessed up to day 100
  Time (days from day 0) to hematopoietic reconstitution (ANC>500/µl, PLT>20000/µl and PLT>50000/µl)
Time to transfusion independence | From date of transplantation (day 0) until the date of first documented transfusion independence, assessed up to day 100
  Time (days from day 0) to transfusion independence
Best disease response within the first 100 days (± 7) after transplantation | Transplantation to day 100 (± 7) after transplantation
  Best disease response within the first 100 days (± 7) after transplantation (according to IWG-criteria for MDS and ELN-criteria for AML)
Disease response and donor chimerism at day +30 (± 3), +60 (± 7) and +100 (± 7) after transplantation | Transplantation until days +30 (± 3), +60 (± 7) and +100 (± 7) after transplantation
  Disease response and donor chimerism at day +30 (± 3), +60 (± 7) and +100 (± 7) after transplantation (according to IWG-criteria for MDS and ELN-criteria for AML)
Time to complete donor chimerism in blood and marrow | From date of transplantation (day 0) until the date of first documented donor chimerism in blood and marrow, assessed up to day 100
  Time (days from day 0) to complete donor chimerism in blood and marrow
Disappearance of molecular markers of disease | From date of transplantation (day 0) until the date of first documented disappearance of individual molecular marker, assessed through study completion, an average of 2 years
  Disappearance of individual molecular markers of disease (time in days from day 0)
Event-free survival | inclusion until 2 years after transplantation
  Event-free survival (death,relapse and disease progression will be recorded as event)
Cumulative incidence of relapse | inclusion until 2 years after transplantation
  Cumulative incidence of relapse (disease progression and relapse will be recorded as event)
Overall survival | inclusion until 2 years after transplantation
  Overall survival (OS, death will be recorded as event)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Kobbe, Prof. Dr., Principal Investigator — Coordinating Investigator
Locations (6):
- Germany (6):
  - Universitätsklinikum Aachen - Med. Klinik IV, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf - Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Köln Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Frankfurt Medizinische Klinik II, Frankfurt
  - Universitätsklinikum Jena - Klinik für Innere Medizin II, Jena
  - Klinikum rechts der Isar der TU München Klinik und Poliklinik für Innere Medizin III, München

IPD SHARING:
Plan to Share IPD: No